CLINICAL TRIAL: NCT05385835
Title: Comparison of Knowledge and Skills Levels of Nurses Who Take Training on Blood Pressure Measurement From The Brachial Artery, After and Before Training
Brief Title: Brachial Artery Blood Pressure Measurement Training
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Burcin Gonenc, Clinical Nurse, Karadeniz Technical University
Other Study IDs: KaradenizTeknikU
Record Dates: First submitted 2022-05-08; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Nurse Training
Keywords: education, nurse, blood pressure measurement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1Nurses: The research is a pre-post-test observation study without a control group, aiming to determine the effect of the training given to nurses on the knowledge and practices of brachial artery blood pressure measurement.
  The research is carried out with a group of 60 nurses.
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — A training module was prepared by explaining the theoretical and practical parts of the application of blood pressure measurement from the brachial artery with a slide presentation and an animation video. The knowledge and skills of nurses in blood pressure measurement before education were measured. The training module was delivered to the nurses from the online system. At the end of the two-week training period, the knowledge and skill levels of the nurses will be measured again.

SUMMARY:
The research is a pre-post-test observation study without a control group, aiming to determine the effect of the training given to nurses on the knowledge and practices of brachial artery blood pressure measurement.

DETAILED DESCRIPTION:
The nurses who were informed about the study and agreed to participate in the study will be followed by two observers at the same time and filled in the "Blood Pressure Measurement Observation Form". Nurses will not be informed by whom and when they will be observed. Each observer will observe each nurse three times (1st observation). After the first observation is over, the "Blood Pressure Knowledge Test" will be applied to the nurses (Pre-test). Then, the training program prepared by the researcher will be uploaded to the hospital automation system and nurses will be asked to follow it. In addition, nurses will be able to log in to the training module and watch the video again and again whenever they want. Nurses will be given a two-week period to follow the training module. At the end of two weeks, the nurses will fill out the "Blood Pressure Information Test" again (2nd test). The "Blood Pressure Measurement Observation Form" will be filled in by the researcher during the blood pressure measurement of the nurses again in the form of the final follow-up (2nd observation).

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Measurement of blood pressure from the brachial artery with a sphygmomanometer
* Caring for adult patients

Exclusion Criteria:

* Using only digital sphygmomanometer in the clinic
* Caring for pediatric patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Nurses working at Kaçkar State Hospital
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
1. The effect of the training given to nurses on the level of knowledge of blood pressure measurement from the brachial artery | About 45 days until 10 June 2022
  The knowledge test prepared consists of 20 questions, each with five options. The achievement test was evaluated by three faculty members who are experts in the field of Nursing Fundamentals. At the same time, the opinions of an expert lecturer in the Department of Measurement and Evaluation in Education were received regarding the achievement test. The experts evaluated all questions on a 4-point Likert scale (1: the item is not suitable, 2: the item should be seriously reviewed, 3: the item should be slightly revised, 4: appropriate). Content validity index (CGI) was calculated according to the evaluations of the experts. It was found sufficient in terms of questions in the achievement test and CGI (CGI min. 0.666, max. 1,000). Knowledge test will be applied to nurses before and after the training.

SECONDARY OUTCOMES:
2. The effect of training given to nurses on brachial artery blood pressure measurement practices | About 45 days until 10 June 2022
  The observation form includes a total of 31 observation steps as "observed (true-false)" and "not observed" in the preparation of the individual and the environment, determination of the appropriate position, selection of the cuff, measurement technique and recording in the application of blood pressure measurement. The observation form was evaluated by three faculty members who are experts in the field of nursing principles. The experts evaluated all questions on a 4-point Likert scale (1: the item is not suitable, 2: the item should be seriously reviewed, 3: the item should be slightly revised, 4: appropriate). Nurses will be observed three times by two observers while measuring blood pressure before and after the training. Kappa analysis and correlation analysis were applied to determine consistency among observers. The minimum Kappa value was obtained as 0.634. A Kappa value between 0.61-0.80 indicates a significant agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Burçin Gönenç, Principal Investigator — KARADENİZ TEKNİK ÜNİVERSİTESİ
Locations (1):
- Karadeniz Teknik Üniversitesi, Trabzon, Turkey (Türkiye)